CLINICAL TRIAL: NCT04202848
Title: The Clinical Study of Modern Therapies on Flora in Body Fluids and Blood of Malignant Tumor Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PJ-KS-KY-2019-134
Record Dates: First submitted 2019-12-08; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer; Breast Cancer; Gastrointestinal Cancer; Malignant Neoplasms
Keywords: Flora
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Gastrointestinal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces, urine, pharyngeal swab specimens from patients with malignant tumors and discarded blood from clinical laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flora analysis — diversity and abundance of bacteria in patients who received malignant tumors

SUMMARY:
The clinical study of modern therapies on flora changing in blood, oral cavity, urethra and intestinal tract of patients with malignant tumors. The study is observational. Patients are diagnosed cancer based on pathology or cell biology. The sample of flora will be obtained from their blood, oral cavity, urethra and intestinal tract, mainly to study what modern therapies lead to the influence of microecological environment including diversity and abundance of bacteria in patients who received malignant tumors. Immunological examination and Blood biochemistry evaluation include the number ratio, activity and function of immune cell, the immune cell marker(CD3, CD4, CD8, etc), C-reactive protein(CRP), tumor necrosis factor(TNF), Inflammatory stimulant factor(IL-2, IL-6, etc), tumor marker(CEA, AFP, etc),etc. Clinical evaluation includes image data(CT/MRI), quality of life(QOL), no disease progression survival, total survival, objective disease remission rate, etc.

DETAILED DESCRIPTION:
This study collected samples of feces, urine, discarded blood and pharyngeal swab specimens from clinical laboratory from patients with malignant tumors in thoracic surgery department, general surgery department, oncology department and etc before and after treatments which contain chemotherapy, radiation therapy, immune targeted, endocrine therapy, surgery, traditional Chinese medicine and other modern therapies. Researchers will analyze the samples by oral flora, urethra, blood flora bacteria, the species diversity and abundance of the intestinal flora. Besides, quantitative analysis of inflammatory stimulators, c-reactive protein and tumor necrosis factor in peripheral blood was conducted to observe the relationship between the change characteristics of blood, oral, intestinal, urinary tract flora and urine composition caused by treatment and the therapeutic effect and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old, male or female
2. Clinical diagnosis of malignant tumors
3. It is planned to receive cancer treatment
4. The genre of therapies is not limited, which contain chemotherapy, radiation therapy, immune targeted, endocrine therapy, surgery, traditional Chinese medicine and other modern therapies

Exclusion Criteria:

1. Cancer treatment before therapies
2. Previous history: He has suffered from intestinal microecology-related diseases such as cirrhosis, ulcerative colitis, Crohn's disease, irritable bowel syndrome, and urinary system diseases
3. Neurological, psychiatric or unconscious disorders.
4. The following drugs were used within 2 weeks before enrollment:

   1. Probiotic preparations, various prebiotic preparations, etc
   2. gastrointestinal peristaltic drug;
   3. Take drugs known to have a significant effect on the intestinal and urethral flora within half a year (such as proton pump inhibitors, purgatives, bismuth, adsorbents, non-steroidal anti-inflammatory drugs, etc.)
5. Other situations that the researcher considers unsuitable to participate in the experiment;

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with malignant tumors
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2022-11-11 (Estimated); Study Completion 2022-11-11 (Estimated)

PRIMARY OUTCOMES:
The change of diversity of intestinal flora in faeces during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of diversity of urethral flora in urine during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of diversity of oral flora in pharyngeal swab during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of diversity of flora in blood during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of abundance of intestinal flora in faeces during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of abundance of urethral flora in urine during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of abundance of oral flora in pharyngeal swab in urine during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of abundance of flora in blood during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of concentration of purine metabolites in urine during therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of concentration of P-hydroxyphenylalanine metabolites in urine | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months

SECONDARY OUTCOMES:
The change of the number of tumor necrosis factor(TNF)-α in blood during the therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of the number of immune cell marker(CD3, CD4, CD8, etc) in blood during the therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of the number of C-reactive protein(CRP) in blood during the therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of the number of tumor marker(CEA, AFP, etc) in blood during the therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months
The change of the number of Gastrin in blood during the therapy | the 1st day before the start of each kind of therapies, through cancer treatment, day 1, day 3, day 7 after treatment completion, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China